CLINICAL TRIAL: NCT02494427
Title: Medico-economic Comparative Assessment of Conventional and CAD/CAM Dental Restorations; Impact on Hospital Dentistry Departments
Brief Title: Comparison of Conventional and CAD/CAM Dental Restorations
Acronym: EVACFAOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K110104
Record Dates: First submitted 2015-06-10; First posted 2015-07-10 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Dental Caries; Tooth Fractures; Tooth Resorption
Keywords: Crowns; Inlays; Onlays
MeSH Terms: conditions — Dental Caries; Tooth Fractures; Tooth Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CAD/CAM manufactured fixed unitary dental prostheses
  Interventions: Device: CAD/CAM manufactured fixed unitary dental prostheses
- 2 (Active Comparator): Conventionally manufactured unitary dental prostheses
  Interventions: Device: Conventionally manufactured unitary dental prostheses

INTERVENTIONS:
Device: CAD/CAM manufactured fixed unitary dental prostheses
  Arms: 1
Device: Conventionally manufactured unitary dental prostheses
  Arms: 2

SUMMARY:
Dental restorations (crowns, inlays or onlays) can be made conventionally or by CAD/CAM. The current literature is weak and does not separate the medical results of these two techniques. However, the efficiencies enabled by CAD/CAM could, for the price of an initial investment, improve service to the patient by reducing the time required for these restorations, and possibly lower care costs.

The aim of the study is to compare immediate medical results and short-term prosthetic restorations made conventionally or by CAD/CAM in randomized patients, and evaluate economic impacts and organizational aspects.

DETAILED DESCRIPTION:
The medico-economic objective of this study is to assess an organizational innovation for patients treated at the hospital for dental substance loss. The intervention study is the availability of such information for the management of patients, not that of its systematic use.

The economic evaluation of this innovation consists of several parts:

1. A costing study seeking to determine the costs of compensation for dental substance loss by conventional technique and CAD/CAM per patient ;
2. Evaluate the cost from an hospital perspective to substitute CAD/CAM to conventional dental treatment equipments;
3. To built a cost-effectiveness ratio comparing the conventional technique and the CAD/CAM on the criterion of proportions of effective restorations obtained .

Assess the medical and medico-technical impact of prosthesis availability from CAD/CAM:

Modifications of treatment plans (some indications of plastic fillings could shift toward CD/CAM restorations?) and/or their chronology (order of execution phases).

The patient cohort is cared for in a hospital Department of Dentistry for oral rehabilitation.

There is indication of at least a partial or total dental crown restoration either by conventional methods or by CAD/CAM (equipoise).

Directly assessable elements are:

at the individual restoration level: Effective restoration time between indication and effective restoration, quality of the restoration, number of clinical sessions required, unitary cost of the restoration at the patient level: compliance, overall duration of treatment, duration of the restoration phase, number of clinical sessions (global and restoration phase) , criteria of quality of life (OHIP, SF36), treatment costs (global and restoration phase) at the hospital level: number of patients cared for per unit of time, number of restorations, revenues, expenses

Patients seeking dental restorations in one of the study centers an needing at least one fixed restoration feasible either by CAD/CAM or conventional means will be selected during their first consultation (excluding emergency consultations). Quality of life (QOL) indices are then recorded.

Two treatment plans are then created, one using conventional means and another using CAD/CAM means as required ; those two plans may differ in steps order. The last treatment step where these plans are identical is the randomization point.

The treatment plans are maintained during the pre-prosthetic phases of the treatment, and updated in case of intercurrent events.

The patient is formally included at the randomization point, and the plan selected by the randomization is carried out. The resource consumptions entailed by the prosthetic steps are recorded.

At the end of treatment, patient satisfaction and QOL indices are recorded. An identical record is made 6 months after the end of treatment.

Further long-term follow-up of the patients included in this study is planned, but will be the object of another protocol.

ELIGIBILITY:
Inclusion criteria :

* The patient is cared for in a hospital department of Dentistry for oral rehabilitation.
* The patient has a dental insurance plan
* There is indication of at least a partial or total dental crown, either by conventional methods or by CAD/CAM ( equipoise clause) .
* It is possible to follow the patient for at least 6 months ( mid-term outcome evaluation beyond the immediate outcome)
* Assessment of the patient to this monitoring (formal informed consent is not required by French law for accepted procedures)

Exclusion criteria :

* mental , linguistic or legal impossibility of understanding the protocol or no consent to participation.
* Follow-up impossible or doubtful
* Contraindication whatsoever to any therapeutic that can be implemented:

  * bruxism and occlusion disorders requiring treatment ( mechanical stresses , ceramic contra-indicated )
  * TMJ disorder (severe limitation of therapeutic options before resolution)
  * known intolerance to a dental material used in the study
* Patients participating in another clinical trial that may have an impact on the oro-facial region (consultation with investigators in the other trial is required before selection and inclusion).

Teeth:

* Need for further prosthetic development (e. g. telescopic milled crown ) .
* Extensive coronary reconstruction requiring de novo root anchorage (post-and-core)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
efficiency (derived from differences in efficacy, safety and costs) | 18 months
  Differential efficiency (derived from differences in efficacy, safety and costs) at end of treatment.

SECONDARY OUTCOMES:
observance (number of visits/number of necessary visits for treatment) | 18 months
  number of visits/number of necessary visits for treatment
patient satisfaction on the VAS scale | 18 months
quality of life measured by SF36 | 18 months
quality of life measured by OHIP14 | 18 months
occurrence of adverse effects | 18 months
Costs | 18 months
  Number of prosthetic treatment sessions + Total prosthetic sessions durations + Medical personal cost + Disposable or semi-disposable consumables + Hospital revenues (as recorded in hospital records)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Azerad, DDS, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service d'Odontologie Hôpital Pitié salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No